CLINICAL TRIAL: NCT06898112
Title: Mixed-methods Protocol for the WiSSPr Study: Women in Sex Work, Stigma and Psychosocial Barriers to Pre-exposure Prophylaxis in Zambia
Brief Title: Mixed-methods Protocol for the WiSSPr Study
Acronym: WiSSPr
Status: Completed | Type: Observational
Sponsor: Centre for Infectious Disease Research in Zambia (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH); University of Washington (Other)
Responsible Party: Sponsor
Other Study IDs: UJMT Fogarty Fellowship 2023; D43TW009340 (NIH)
Record Dates: First submitted 2025-03-11; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: PrEP Uptake
Keywords: stigma; prep; sex work; women; zambia; southern africa; community-based participatory research; community advisory board
MeSH Terms: conditions — Social Stigma; Sex Work

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- PrEP initiators: women who initiate on PrEP
  Interventions: Drug: PrEP
- PrEP refusers: women who refuse PrEP

INTERVENTIONS:
Drug: PrEP — oral PrEP
  Groups: PrEP initiators

SUMMARY:
WiSSPr is a prospective observational cohort study grounded in community-based participatory research principles with a community advisory board (CAB) of key population (KP) civil society organi sations (KP-CSOs) and the Ministry of Health (MoH).

DETAILED DESCRIPTION:
WiSSPr is a prospective observational cohort study grounded in community-based participatory research principles with a community advisory board (CAB) of key population (KP) civil society organi sations (KP-CSOs) and the Ministry of Health (MoH). We will administer a one-time psychosocial survey vetted by the CAB and follow 300 WESW in the electronic medical record for three months to measure PrEP initiation (#/% ever taking PrEP) and persistence (immediate discontinuation and a medication possession ratio). We will conduct in-depth interviews with a purposive sample of 18 women, including 12 WESW and 6 peer navigators who support routine HIV screening and PrEP delivery, in two community hubs serving KPs since October 2021. We seek to value KP communities as equal contributors to the knowledge production process by actively engaging KP-CSOs throughout the research process. Expected outcomes include quantitative measures of PrEP initiation and persistence among WESW, and qualitative insights into the enablers and barriers to PrEP use informed by participants' lived experiences. https://doi.org/10.1136/bmjopen-2023-080218

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria: (1) identify as a cis-gendered or transgendered woman, (2) age ≥ 18 years, (3) earns a significant amount of income from exchanging sex for money or goods in the last 3 months, (4) HIV-negative status and eligible for PrEP according to national guidelines, (5) not planning to transfer care to another site within the next 30 days, (6) speaks English or ChiNyanja or IchiBemba and (7) willing and able to provide written informed consent

Exclusion Criteria:

* Exclusion criteria: (1) do not identify as a woman, (2) age < 18 years old, (3) has not earned a significant amount of income from exchanging sex for money or goods or has earned for < 3 months, (4) HIV-positive status or status is unknown or ineligible for PrEP, (5) planning to transfer care to another site within the next 30 days, (6) unable to speak English or ChiNyanja or IchiBemba and (7) not willing or able to provide written informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — cis or trans-gender women self identified
Study Population: The study population is composed of adult WESW who are living or working within the catchment areas of two community hubs located within urban Lusaka. Based on CIDRZ's prior published work, we anticipate that the study population will be comprised largely (63%) of younger women (18 - 29 years old).
Sampling Method: Non-Probability Sample
Enrollment: 299 (Actual)
Dates: Start 2023-07-18 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
PrEP initiation (#/% ever taken PrEP) | 3 months
  PrEP initiation (Number or percentage of Women Engaging in Sex Work (WESW) initiating on PrEP)
PrEP Persistence (#/ % eligible refills obtained until first discontinuation) | 3 months
  PrEP persistence. Number or percentage of women engaging in sex work with high levels of stigma who will persist on PrEP

CONTACTS AND LOCATIONS:
Overall Officials: Ramya Kumar, PhD, MPH, Principal Investigator — University of Washington
Locations (1):
- Centre for Infectious Disease Research Zambia, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: No
Vulnerable population of sex workers in a country where sex work is largely criminalized, and there is a risk of harm if the data is identifiable even with common identifiers like name is removed.

REFERENCES:
- See also: Protocol paper — https://bmjopen.bmj.com/content/14/9/e080218